CLINICAL TRIAL: NCT02718066
Title: A Phase 1b/2 Study to Assess the Safety and Efficacy of HBI-8000 in Combination With Nivolumab in Subjects With Advanced Solid Tumors Including Melanoma, Renal Cell Carcinoma (RCC), and Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of HBI-8000 With Nivolumab in Melanoma, Renal Cell Carcinoma and Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-8000-302
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Melanoma; Renal Cell Carcinoma; Non-Small Cell Lung Cancer
Keywords: HBI-8000; Nivolumab; Melanoma; Renal Cell Carcinoma; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — HBI-8000; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HBI-8000 in combination with nivolumab (Experimental): HBI-8000 dose escalation 20mg, 30mg, 40mg, orally, twice weekly; in combination with Nivolumab 240mg intravenous infusions every 2 weeks for Phase 1b and in accordance with the manufacturer package insert and institution's prescribing practice for Phase 2.
  Interventions: Drug: HBI-8000 in combination with nivolumab

INTERVENTIONS:
Drug: HBI-8000 in combination with nivolumab — Phase 1b: HBI-8000, orally, twice a week, dose escalation 20mg, 30mg, 40mg; in combination with nivolumab 240mg intravenous infusion every 2 weeks.
  Phase 2: HBI-8000 MTD or 40mg; in combination with nivolumab in accordance with the manufacturer package insert and institution's prescribing practice.
  Other Names: For HBI-8000: Chidamide, CS055; for nivolumab: OPDIVO

SUMMARY:
A Phase 1b/2 Study to Assess the Safety and Efficacy of HBI-8000 in Combination with Nivolumab in Patients with Advanced Solid Tumors Including Melanoma, Renal Cell Carcinoma (RCC), and Non-Small Cell Lung Cancer (NSCLC).

The primary objective of this study is:

-To evaluate the safety and tolerability of HBI-8000 when combined with a standard dose and regimen of nivolumab, and to evaluate frequency and severity of toxicities of this combination treatment

The secondary objectives of this study include:

* To explore the efficacy of study treatment as measured by Objective Response Rate (ORR), Disease Control Rate (DCR), Clinical Benefit Rate (CBR), Duration of Response (DoR), Progression-Free Survival (PFS) in all subjects treated at RP2D
* To obtain pharmacokinetics of twice weekly HBI-8000 when administered in combination with nivolumab administered once every two weeks (Phase 1b all sites)
* To obtain pharmacokinetics of twice weekly HBI-8000 when administered in combination with nivolumab administered per package insert dose and administration (Phase 2 selected sites)
* To characterize the effect of HBI-8000 on the electrocardiogram QT corrected (QTc) interval (Phase 1b only)

Exploratory:

* To investigate the kinetics and extent of histone acetylation in peripheral blood mononuclear cells (PBMC) at the RP2D of HBI-8000 (Phase 2 only)
* To explore potential biomarkers for disease response through sequential sampling of blood and/or tumor tissue in subjects consenting to correlative sub-studies at participating sites (Phase 2 only)

Dose Escalation (Phase 1b) will include up to 18 subjects, followed by Cohort Expansion (Phase 2) including up to 100 subjects (melanoma up to 60 subjects and NSCLC up to 40 subjects at MTD and/or RP2D.

DETAILED DESCRIPTION:
A Phase 1b/2 Study to Assess the Safety and Efficacy of HBI-8000 in Combination with Nivolumab in Patients with Advanced Solid Tumors Including Melanoma, Renal Cell Carcinoma (RCC), and Non-Small Cell Lung Cancer (NSCLC).

The primary objective of this study is:

-To evaluate the safety and tolerability of HBI-8000 when combined with a standard dose and regimen of nivolumab, to determine Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) and to evaluate frequency and severity of toxicities of this combination treatment

The secondary objectives of this study include:

* To explore the efficacy of study treatment as measured by Objective Response Rate (ORR), Disease Control Rate (DCR), Clinical Benefit Rate (CBR), Duration of Response (DoR), Progression-Free Survival (PFS) in all subjects treated at RP2D
* To obtain pharmacokinetics of twice weekly HBI-8000 when administered in combination with nivolumab administered once every two weeks (Phase 1b all sites; Phase 2 selected sites)
* To characterize the effect of HBI-8000 on the electrocardiogram QT corrected (QTc) interval (Phase 1b only)

Exploratory:

-To investigate the kinetics and extent of histone acetylation in peripheral blood mononuclear cells (PBMC) at the RP2D of HBI-8000 (Phase 2 only)

Dose Escalation (Phase 1b) will include up to 18 subjects, followed by Cohort Expansion (Phase 2) including up to 100 subjects (melanoma up to 60 subjects and NSCLC up to 40 subjects) at MTD and/or RP2D.

HBI-8000 tablets will be administered at 20, 30, 40 mg/dose, orally twice a week until MTD or 40 mg in Phase 2, if MTD is not reached.

Nivolumab: 240 mg intravenous infusions every 2 weeks for Phase 1b and in accordance with the manufacturer package insert and institution's prescribing practice for Phase 2.

A treatment cycle consists of 28 days. Treatment continues until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria. Patients may be entered in the study only if they meet all of the following criteria:

1. Adults at least 18 years of age. 2. Eastern Cooperative Oncology Group (ECOG) performance status ≤1. 3.

1. Subjects with histopathologically or cytologically confirmed diagnosis of non-uveal Melanoma, RCC or NSCLC, for whom the use of nivolumab is indicated. NSCLC subjects with EGFR or ALK genomic aberrations in tumor should have disease progression on FDA-approved therapy for these aberrations prior to receiving nivolumab (Phase 1b).
2. Subjects with histopathologically or cytologically confirmed diagnosis of non-uveal Melanoma, or NSCLC, for whom the use of nivolumab is indicated. With Protocol Amendment 5, subjects with NSCLC are not eligible for enrollment.
3. Non-uveal melanoma and NSCLC patients whose disease has progressed after achieving SD for at least 3 months, PR or CR as the best response that has been documented by imaging studies (Phase 2 expansion).With Protocol Amendment 5, subjects with NSCLC are not eligible for enrollment.

   4. Subject must have at least one measurable target lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1. Melanoma subjects participating in the optional serial tumor biopsy sub-study must have tumor tissue available from a metastatic or unresectable site for PD-L1 and correlative biomarker analysis.

   5. All prior systemic therapy (chemotherapy, mutation targeting therapy, immune checkpoint therapy), surgical or radiation treatment must have been completed at least 4 weeks before study drug administration (2 weeks for palliative radiotherapy, 1 week for minor surgery) pending full recovery from therapy.

   6. The following laboratory results within 7 days prior to study drug administration: Adequate hematopoietic, electrolyte, hepatic, and renal laboratory findings as defined below: WBC ≥3000/μL, Neutrophils ≥1500/μL, Platelets ≥100x103/μL, Hemoglobin ≥9.0g/dL independent of transfusion, Creatinine ≤1.5mg/dL, AST and ALT ≤3x ULN, Alkaline phosphatase ≤2.5x ULN unless bone metastases present, Bilirubin ≤1.5x ULN (unless known Gilbert's disease where it must be ≤3x ULN) and serum albumin ≥3.0g/dL.

   7. Life expectancy ≥12 weeks. 8. A negative serum pregnancy test at baseline for women of childbearing potential.

   9. Are willing to abstain from heterosexual activity or practice physical barrier contraception prior to time of study entry to at least 5 months after the last day of treatment.

   10. Have the ability to understand and the willingness to sign a written informed consent document.

   Exclusion criteria. Subjects who fulfill any of the following criteria at screening will not be eligible for admission into the study:
   1. History of Grade 3 or above hypersensitivity reactions to other monoclonal antibodies.
   2. Subjects with a history of a cardiovascular illness including: congestive heart failure (New York Heart Association Grade III or IV); unstable angina or myocardial infarction within the previous 6 months; or symptomatic cardiac arrhythmia despite medical management.
   3. Uncontrolled hypertension, SBP >160 or DBP >100.
   4. Subjects with active brain metastasis; previously treated brain metastasis is allowed if it has been stable for 4 weeks or more and not requiring steroids.
   5. Presence of leptomeningeal disease.
   6. History of hemorrhagic diarrhea, inflammatory bowel disease, active uncontrolled peptic ulcer disease or recurrent pleural effusion requiring repetitive palliative thoracentesis within 3 months prior to study entry, except for subjects with a pleurex port. and immune-mediated toxicity leading to treatment discontinuation
   7. Active, known, or suspected autoimmune disease, except for type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia).
   8. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
   9. Known history of testing positive for human immunodeficiency virus (HIV), known acquired immunodeficiency syndrome (AIDS).
   10. Active hepatitis B (serum hepatitis B surface antigen [HBV sAg] positive), or hepatitis C (HCV antibody test or serum hepatitis C RNA positive) indicating acute or chronic infection.
   11. Subjects with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted.
   12. Use of other investigational agent (drug not marketed for any indication) within 28 days or at least 5 half-lives (whichever is shorter) before study drug administration.
   13. Pregnant or breast-feeding women.
   14. Second malignancy unless in remission for 2 years, except for non-melanomatous skin cancer, carcinoma in situ of the cervix treated with curative intent, curatively treated prostate cancer with prostate-specific antigen (PSA) <0.1 ng/mL.
   15. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events.
   16. Unwilling or unable to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Determination of the Recommended for Phase 2 Dose (RP2D) (mg) | 12 months
  Determination of the Recommended for Phase 2 Dose (RP2D) (mg)

SECONDARY OUTCOMES:
Efficacy Outcome: Response Rate (%). | 18 months
  Objective Response Rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil I Khushalani, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, FL
Locations (6):
- United States (6):
  - [Site 02] Mayo Clinic Arizona, Phoenix, Arizona
  - [Site 11] University of California, San Diego Medical Center, La Jolla, California
  - [Site 01] Hematology - Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - [Site 09] H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida
  - [Site 13] Frederick Memorial Hospital d/b/a James M Stockman Cancer Institute, Frederick, Maryland
  - [Site 12] University of Texas M.D. Anderson Cancer Center - Investigational Cancer Therapeutics, Houston, Texas

IPD SHARING:
Plan to Share IPD: No